CLINICAL TRIAL: NCT01320592
Title: A Phase 1 Trial of PD0332991 and Paclitaxel in Patients With Rb-Expressing Advanced Breast Cancer
Brief Title: PD0332991/Paclitaxel in Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 02111
Record Dates: First submitted 2011-03-16; First posted 2011-03-22 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
Keywords: Patient must have histologically or cytologically-confirmed metastatic; breast cancer; Any ER, PR or Her2 status is allowed.; Tumor must express Retinoblastoma (Rb) protein, defined as; any measurable staining by immunohistochemistry on the invasive tumor component; <3 prior cytoxic chemotherapy regimens for metastatic disease.; Performance status of 0-1 on the Eastern Cooperative Oncology Group Performance Scale and life expectancy > 3 months.; Patient must have evaluable disease. Measureable disease is not required.; The subject has adequate organ function
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PD0332991 and Paclitaxel (Experimental): PD0332991 in combination with weekly paclitaxel at a fixed dose of 80 mg/m2
  Interventions: Drug: PD0332991; Drug: Paclitaxel

INTERVENTIONS:
Drug: PD0332991
Drug: Paclitaxel

SUMMARY:
This study is a phase I, single arm, open-label trial of PD0332991 in combination with Paclitaxel in patients with Rb-expressing metastatic breast cancer. Up to 20 patients are anticipated to be enrolled to reach the Maximum Tolerated Dose (MTD) of PD0332991 in combination with Paclitaxel. Once the MTD is established, an additional expanded cohort of 10 patients will be enrolled at that dose to establish the Recommended Phase 2 Dose (RP2D), obtain additional safety data and perform exploratory biomarker studies.

DETAILED DESCRIPTION:
This study is a phase I, single arm, open-label trial of PD0332991 in combination with paclitaxel in patients with Rb-expressing metastatic breast cancer. Patients will be treated as shown in the schema below. Up to 20 patients are anticipated to be enrolled to reach the MTD of PD0332991 in combination with Paclitaxel. Once the MTD is established, an additional expanded cohort of 10 patients will be enrolled at that dose to establish the RP2D, obtain additional safety data and perform exploratory biomarker studies. The primary endpoint will be assessed after one cycle of therapy. Patients will remain on study until dose limiting toxicity, disease progression or physician/patient discretion. Safety assessment will continue for the duration of patient participation.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have histologically or cytologically-confirmed metastatic breast cancer. Any ER, PR or Her2 status is allowed.
* Tumor must express Retinoblastoma (Rb) protein, as defined as any measureable staining by immunohistochemistry
* Male or female and > 18 years of age on the day of signing informed consent.
* Patient must have received < prior cytotoxic regimens for metastatic breast cancer. This does not include cytoxic regimens used in the adjuvant setting.
* Performance status of 0-1 on the Eastern Cooperative Oncology Group Performance Scale and life expectancy > 3 months.
* patient on the dose-escalation portion of the trial must have evaluable disease, defined as either measurable (by RECIST) or non-measurable disease (e.g. bone mets, pleural effusion or lymphangitic spread). Measurable disease is required for patients in the expanded RP2D cohort.
* The subject must have adequate organ function, defined as follows:

Bilirubin < 1.5 x upper normal limit or calculated creatinine clearance > 60 mL/min, and for subjects without liver metastases: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x upper normal limit

* For subjects without extensive bone metastases: alkaline phosphatase levels < 2.5 x upper normal limit .
* For subjects with extensive bone metastases: alkaline phosphatase levels < 5 x upper normal limit .
* The subject must have adequate marrow function, defined as follows
* Absolute neutrophil count (ANC) >1500/mm
* Platelets > 100,000/mm
* Hemoglobin > 9 g/dL
* Female patient of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to receiving the first dose of study medication and agree to the use of effective methods of contraception while on study.
* Patient must be capable of, and must voluntarily agree to participate by giving written informed consent.
* Patient must be able to swallow capsules and has no surgical or anatomical condition that will preclude the patient from swallowing and absorbing oral medications on an ongoing basis.
* Prior taxane therapy in the adjuvant or metastatic setting is allowed.
* Concomitant use of biphosphonates is allowed.
* Patients with stable, treated CNS disease are eligible.

Exclusion Criteria:

* Patient who has had chemotherapy, radiotherapy or hormonal therapy within 3 weeks (6 weeks for nitrosoureas, mitomycin C or bevacizumab), or who has not recovered from the adverse events due to previous agents administered more than 4 weeks prior to Study Day 1. If the patient has residual toxicity from prior treatment, toxicity must be < Grade 1.
* patients less than 4 weeks post major surgical procedure (all surgical wounds must be fully healed). For the purpose of this criterion, a major surgical procedure is defined as one requiring the administration of general anesthesia.
* Patient has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. However, patients with CNS metastases (including brain metastases) who have completed a course of radiotherapy are eligible for the study provided they are clinically stable. Oral corticosteroids for control of CNS symptoms are allowed.
* Patient has known hypersensitivity to the components of study drug or its analogs.
* The subject has uncontrolled intercurrent illness including, but not limited to Ongoing or active infection
* Diabetes mellitus
* Hypertension
* Symptomatic congestive heart failure, unstable angina pectoris, stroke or myocardial infarction within 3 months.
* Patient has baseline neuropathy of > grade 2
* Patients who have known allergic reactions to Paclitaxel or IV Contrast Dye despite standard prophylaxis.
* The subject is pregnant or breastfeeding
* The subject is known to be positive for the human immunodeficiency virus (HIV). Note: baseline HIV screening is not required.
* The subject is unable eor unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
To Determine the Adverse Events of PD0332991 | weekly paclitaxel at a fixed dose of 80 mg/m2 and to assess the safety of the combination after 3 cycles of therapy (cycles are 28 days) .
  To determine the maximally-tolerated dose and safety of PD0332991 in combination with a fixed, weekly dose of Paclitaxel of 80 mg/m2 and to characterize the safety of the combination during the first three cycles of therapy.

SECONDARY OUTCOMES:
Maximally Tolerated Dose in an expanded Cohort of Breast Cancer Patients | weekly paclitaxel at a fixed dose of 80 mg/m2 and to assess the safety of the combination after 3 cycles of therapy (cycles are 28 days)
  To explore the activity of the combination at the MTD in an expanded cohort of breast cancer patients.
To explore the relationship between selected biomarkers and efficacy, tolerability and safety outcomes | weekly paclitaxel at a fixed dose of 80 mg/m2 and to assess the safety of the combination after 3 cycles of therapy (cycles are 28 days)
  To explore the relationship between selected biomarkers and efficacy, tolerability and safety outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Clark AS, McAndrew NP, Troxel A, Feldman M, Lal P, Rosen M, Burrell J, Redlinger C, Gallagher M, Bradbury AR, Domchek SM, Fox KR, O'Dwyer PJ, DeMichele AM. Combination Paclitaxel and Palbociclib: Results of a Phase I Trial in Advanced Breast Cancer. Clin Cancer Res. 2019 Apr 1;25(7):2072-2079. doi: 10.1158/1078-0432.CCR-18-0790. Epub 2019 Jan 11. PMID 30635336